CLINICAL TRIAL: NCT00653367
Title: Post Thoracotomy Pain After Nerve Section
Brief Title: Evaluation of Chronic Pain After Nerve Section During Thoracotomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD Kim Wildgaard, Section for Surgical Pathophysiology 4074
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RH-EKPF-2008-01
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2011-08

CONDITIONS: Lung Cancer
Keywords: Thoracotomy; Nerve section; QST; Quantitative Sensory Test; Muscle sparing Posterolateral thoracotomy; Chest; Wall; Surgical; Incision; Tumors or cancer of the lung
MeSH Terms: conditions — Lung Neoplasms; Surgical Wound; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS (Experimental): Nerve section of intercostal nerve during surgery
  Interventions: Procedure: Nerve section
- Control (No Intervention): Control

INTERVENTIONS:
Procedure: Nerve section — Intercostal nerve is divided during surgery
  Arms: NS

SUMMARY:
The purpose of this study is to investigate if controlled nerve section reduces chronic pain after thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients included for anterior or lateral thoracotomy

Exclusion Criteria:

* Unable to give consent due to age, cognitive reduction or otherwise
* Neurological disease or symptoms affection thoracic area
* Chronic pain prior to surgery
* Inability to supply the patient with an epidural catheter
* Pneumonectomy
* Prolonged infection at surgical site
* Invasive tumor growth
* Need for repeated surgery at site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain (NRS) | 3 months postoperatively

SECONDARY OUTCOMES:
QST parameters (sensory thresholds to cool/Warmth) | 3 months postoperatively
Social well-being (HADS / PCS) | 3 months postoperatively
Function (pain impairment of Activities of Daily Life) | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wildgaard, MD, Principal Investigator — Section for Surgical Pathophysiology 4074; Henrik Kehlet, MD, Phd, Pro, Study Chair — Section for Surgical Pathophysiology 4074
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark